CLINICAL TRIAL: NCT02080416
Title: A Pilot Trial of Nelfinavir for the Lytic Activation and Treatment of Gammaherpesvirus-Related Tumors
Brief Title: Nelfinavir for the Treatment of Gammaherpesvirus-Related Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Very slow accrual; terminated to allow resources to be utilized more effectively on other studies. No data analysis completed, nor any conclusions reached.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J13174; NA_00092477 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Non-Hodgkin Lymphoma; Hodgkin Lymphoma; Kaposi Sarcoma; Gastric Cancer; Nasopharyngeal Cancer; EBV; Castleman Disease
Keywords: EBV; KSHV; malignancy; lymphoma; sarcoma; virus-associated
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Sarcoma, Kaposi; Stomach Neoplasms; Nasopharyngeal Neoplasms; Castleman Disease; Neoplasms; Lymphoma; Sarcoma | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir (Experimental): Nelfinavir twice daily on days 1-14 of a 14-day cycle for 4 cycles
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir — Nelfinavir will be given 3000 mg orally twice daily on days 1-14 of a 14-day cycle. NFV will be continued in patients tolerating therapy for 4 cycles (8 weeks).
  Other Names: Viracept®

SUMMARY:
The goals of this study is to determine if nelfinavir can target Epstein-Barr virus (EBV) and Kaposi sarcoma-associated herpesvirus (KSHV) in patients with certain cancers.

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) and Kaposi sarcoma-associated herpesvirus (KSHV) are gammaherpesviruses that are associated with a variety of human cancers, including a subset of lymphomas, carcinomas, and sarcomas. In tumors the virus typically exists in a latent state. In latently infected cells, the vast majority of viral genes are not expressed and there is little to no production of infectious virions. The virus replicates in tandem with cell division using cellular machinery. This highly restricted pattern of gene expression allows the virus to evade immune recognition and clearance.

Currently, the treatment approach to virally-associated malignancies is no different than the treatment approach to the same tumors where there is no viral association. Yet, the presence of virus within these tumors offers an opportunity to develop virus-specific, targeted therapies in these diseases. Such therapies might not only be more effective but also less toxic. EBV- and KSHV-associated cancers are more common in patients with HIV, congenital immunodeficiencies, or other immunosuppression, such as transplant recipients. These patients in particular would benefit from more targeted treatment approaches to their malignancies, potentially sparing the toxicities of cytotoxic chemotherapy in an already immunocompromised patient population.

Activation of lytic gene expression in virally-infected tumors may enhance tumor-specific cell killing through multiple mechanisms. Importantly, the cytotoxic effects of antiviral nucleoside analogues, such as acyclovir and its cogeners, depend on the activity of viral kinases which are only expressed during lytic replication. Because EBV(+) or KSHV(+) tumors are characterized by latent viral infection, these antiviral drugs as a single agent are not active in these tumors. However, if lytic gene expression could be activated in virally-associated tumors, this could render EBV(+) and KSHV(+) tumor cells susceptible to killing by antiviral nucleoside analogues.

Nelfinavir (NFV), an FDA-approved protease inhibitor for the treatment of HIV, has been shown to be a potent activator of lytic gene expression of EBV(+) and KSHV(+) cancer cell lines. Furthermore, NFV is able to activate lytic gene expression of EBV and KSHV at drug levels that are achievable in humans. There is also growing evidence that NFV has antitumor activity.

The goals of this study is to determine if NFV activates lytic gene expression in the tumors and causes tumor regression in patients with EBV(+) or KSHV(+) cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Biopsy proven EBV(+) or KSHV(+) malignancy
* Relapsed/refractory disease failing > 2 prior therapies
* Measurable, non-bony disease (at least one lesion on radiographic or physical exam assessment measuring > 2 cm in longest axis)
* KS patients with skin-only disease must have cutaneous lesions amenable to four 3 mm punch biopsies during the course of the study
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Life expectancy of greater than 12 weeks
* Patients must be able to lie flat for at least 60 minutes and fit on a PET-CT scanner
* Ability to comply with an oral drug regimen
* Females of childbearing potential must have a negative pregnancy test at screening
* Patients must have normal organ and marrow function as defined below within 14 days of study entry

Exclusion Criteria:

* Patients with HIV-associated primary central nervous system lymphoma
* Radiotherapy or chemotherapy ending within 14 days of study enrollment
* Patients currently on other protease inhibitors
* Chronic diarrhea
* Acute, active infection within 14 days of enrollment
* Patients on active treatment for hypo- or hyperthyroidism
* End-stage liver disease unrelated to tumor
* Hepatitis B or hepatitis C infection
* Use of any other type of investigational agent or treatment concurrently or within 28 days before the first dose of study treatment
* History of iodine hypersensitivity
* Females who are pregnant or breastfeeding
* Physical or psychiatric conditions that in the estimation of the investigator place the patient at high risk of toxicity, non-compliance, or inability to complete the study requirements
* Use of drugs to treat or prevent herpesvirus infections
* Essential medication that is known to interact with nelfinavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Lytic activation of viral gene expression by NFV | Day 4 and day 5 of Cycle 1
  To determine if NFV activates lytic gene expression in the tumors of patients with EBV(+) or KSHV(+) cancers, as evidenced by the ability to image the tumor with [124I]fialuridine-PET-CT.

SECONDARY OUTCOMES:
Serial assessment of methylation of viral DNA | Day 4 of Cycle 1, at the end of cycles 1-4, 2 weeks post-treatment, and 4 weeks post-treatment
  The methylation of viral DNA in plasma at baseline and during the course of NFV therapy and follow-up will be determined for each patient.
Serial assessment of viral copy number in plasma | Day 4 of Cycle 1, at the end of cycles 1-4, 2 weeks post-treatment, and 4 weeks post-treatment
  Viral DNA copy number in plasma at baseline and during the course of NFV therapy and follow-up will be determined for each patient by quantitative polymerase chain reaction assay (qPCR).
Tolerability of high-dose nelfinavir | Every week up to 2 weeks post-treatment
  The tolerability of high-dose NFV in patients with relapsed/refractory EBV(+) or KSHV(+) tumors will be determined by evaluation of dose limiting toxicities (DLT).
Tumor regression and response | Within 2 weeks of ending treatment
  The responses of EBV(+) and KSHV(+) tumors after 4 cycles of NFV therapy will be assessed by CT for solid tumors, CT or PET-CT for lymphomas and lymphoproliferative disorders, and skin exam with lesion measurements for KS.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ambinder, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Study terminated; no data analysis completed